CLINICAL TRIAL: NCT02189889
Title: Active Preoperative Anemia Management to Reduce Erythrocyte Transfusion in Patients Undergoing Cardiac Surgery (APART): A Pilot, Feasibility Study
Brief Title: Active Preoperative Anemia Management in Patients Undergoing Cardiac Surgery
Acronym: APART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Initial patients were seen at St Paul Hospital. Enrollment changes occurred with the move to Clements Hospital. We were unable to identify an infusion room at CUH despite an exhaustive search for alternatives and forced to terminate early.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Philip Greilich, MD, FASE, Professor and Holder S.T. "Buddy" Harris Distinguished Chair in Cardiac Anesthesiology, Quality Officer, University of Texas Healthcare System, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APART.V1.2013
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Anemia; Cardiovascular Disease
Keywords: Active preoperative anemia management; Erythrocyte transfusion; RBC transfusion; Red cell transfusion; Transfusion in cardiac surgery; Anemia treatment with erythropoietin; Anemic cardiac surgery patients; Erythrocyte stimulating agent (ESA); Iron deficiency anemia; EPO; Feraheme
MeSH Terms: conditions — Anemia; Cardiovascular Diseases; Anemia, Iron-Deficiency | interventions — Erythropoietin; Ferrosoferric Oxide; ferryl iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO and Feraheme (Active Comparator): Patients in the treatment group will receive a subcutaneous injection of EPO 300U/kg at the Baseline visit, the Preoperative visit and on POD 2; and an infusion of Feraheme 510mg at the Baseline visit and the Preoperative visit.
  Interventions: Drug: EPO; Drug: Feraheme
- Control (No Intervention): The control group will receive no preoperative intervention for anemia. The exception being iron deficiency anemia found during baseline. If laboratory values indicate iron deficiency, oral iron will be recommended to take until surgery.

INTERVENTIONS:
Drug: EPO — The treatment group will receive up to three doses of EPO 300U/kg. The first dose of study medication will be administered up to 28 days before the day of surgery and the second will be administered 1-7 days before the day of surgery. These first two doses will be given at least 7 days apart. A third dose may be administered two days following surgery. All 3 doses will be administered per surveillance strategy guidelines.
  Other Names: erythropoietin
  Arms: EPO and Feraheme
Drug: Feraheme — Supplementation with Feraheme, 510mg delivered as an IV infusion, will be given following the first two preoperative doses of EPO.
  Other Names: IV iron
  Arms: EPO and Feraheme

SUMMARY:
Anemia which is a decreased blood count or lower than normal hemoglobin (hgb), is a major health problem for patients having heart surgery. Hemoglobin is the part of our blood that carries oxygen from the lungs to the rest of the body. Anemia that is present before surgery, called preoperative anemia, is a risk factor for an increased chance of morbidity (illness) and/or mortality (death) after heart surgery. It is also an important indicator of blood transfusion necessity. Recent clinical research investigations done to study preoperative anemia suggest a blood transfusion can damage the immune system (the system that protects us from disease) which can lead to infection, organ dysfunction (especially of the heart, kidney, brain), prolonged hospital stays, as well as increased supplies, resources and cost in surgical patients. Comprehensive anemia management can reduce or eliminate the need for blood transfusions and provide better outcomes after surgery. Therefore, controlling anemia before surgery is extremely important, and could be a lifesaving measure.

This pilot, feasibility study is being done for several reasons. First of all, it will test the the safety and effectiveness of using a short-course of two medications, erythropoietin (EPO) and Feraheme (iron given intravenously [IV]), to increase hemoglobin levels in order to improve preoperative anemia, reduce transfusions and lower postoperative complications in anemic patients undergoing heart surgery. Secondly, findings will be used to design a large randomized controlled trial (RCT). The RCT will establish a protocol to actively manage anemia before surgery, thus reducing transfusions during surgery and improving recovery afterwards. It will also help identify valuable information regarding what needs to be done for timely completion of the planned RCT.

EPO is a medication approved by the Food and Drug Administration (FDA) used to treat anemia in patients with certain conditions in order to reduce blood transfusions. And although approved for use during surgery, it has not been FDA approved for use in cardiac (heart) or vascular (blood vessels, including veins and arteries) surgery. Common side effects include nausea, vomiting, itching, headache, injection site pain, chills, deep vein thrombosis (blood clot), cough, and changes in blood pressure (BP). Feraheme is an iron replacement product approved for the treatment of low iron anemia in adult patients. It may cause serious allergic reactions, including anaphylaxis (severe, whole body allergic reaction), as well as low BP and excessive iron storage.

Patients meeting all eligibility requirements that consent to participate will be randomized into the study. Randomization is being placed by chance (like a flip of a coin) into one of two study groups, the treatment group or the control group. There is an equal chance of being placed into either group, which will be done by a computer.

1. The Treatment Group will receive a 300 unit (U) per kilogram (kg) injection of EPO and a 510 milligram (mg) IV infusion of Feraheme 7-28 days before the day of surgery. And again 1-7 days before the day of surgery, a second dose of both of these medications will be given. The third dose, of EPO only, will be administered 2 days after surgery. Before initiating a dose or giving a subsequent dose, laboratory parameters will be measured to assess the hemoglobin level and response to the medication. If blood values increase too rapidly or are too high, the meds will not be started or, if already dosed, they will not be given again.
2. The Control Group will receive no preoperative intervention for anemia unless lab results show iron deficiency anemia. The control group will be screened for the presence of iron deficiency anemia by evaluating blood laboratory values drawn during the baseline or preoperative visit. If lab results indicate iron deficiency anemia, over-the-counter oral iron will be recommended, to take until the day of surgery. In doing so, patients may benefit by potentially reducing the need for blood transfusions.

Data will be collected from all participants from the preoperative visits throughout the admission, including lab results, medications, vital signs, information about the procedure, transfusions, and any problems or adverse events.

DETAILED DESCRIPTION:
Anemia and transfusion are independent predictors of morbidity and mortality in the cardiac surgical patient population. Even so, active preoperative anemia management is not currently the standard of care at our institution. Cost associated with erythrocyte transfusions at University of Texas Southwestern (UTSW) University Hospitals exceeds twenty million dollars annually, not including costs associated with treatment of known complications of red cell transfusions (renal insufficiency, respiratory failure, infection and prolonged length of stay, etc). Fifty percent of our cardiac surgical population suffer from preoperative anemia and 79% of these patients will receive one or more red blood cell (RBC) transfusions. In contrast, the incidence of RBC transfusion was only 35% in those without preoperative anemia in the calendar year 2011-12.

The mechanism of injury in patients with preoperative anemia is either the duration/intensity of the anemia exposure and resultant organ ischemia, or the harmful effects of erythrocyte transfusion(s) itself. Active preoperative anemia management is a strategy that attempts to minimize both of these events, and in doing so, exert an additive or possibly synergistic effect on improving clinical outcomes. A randomized controlled trial utilizing a standardized transfusion strategy is a necessary step in determining if increases in preoperative hemoglobin lead to improved outcomes. A pilot, feasibility study is the first essential step in insuring the adequacy of future trials designed to answer this important question.

The APART study is being conducted to test the safety and efficacy of using a short-course (1-4 weeks) of EPO plus Feraheme to increase erythrocyte mass. The findings will be used to guide the design of a randomized, controlled trial (RCT) that examines the effects of active preoperative anemia management on erythrocyte transfusion and clinical outcomes. The RCT will test the hypothesis that a short-course (1-4 weeks) of EPO plus Feraheme is superior to the standard of care (SOC) at reducing transfusion and improving outcomes in anemic patients scheduled for cardiac surgery. Means and standard deviations derived from pilot data on changes in hemoglobin levels, reticulocyte counts and differences in erythrocyte transfusions and clinical outcomes will be analyzed for possible use in sample size calculations for the larger RCT. This pilot will also provide information in determining logistics for timely completion of the RCT, and will also address data collection, data management, adherence to the study protocol, transfusion and surveillance strategies and classification of clinical outcomes and adverse events.

Pilot Study Specific Aims Include:

1. To determine the proportion of patients who fulfill all the eligibility criteria for the study and agree to be part of a randomized trial of short-course EPO plus supplemental Feraheme (up to 3 doses given over a 1-4 week interval prior to surgery) vs. standard of care management in patients scheduled for coronary bypass grafting (CABG), valve surgery, or CABG/valve surgery.
2. To determine the adherence of patients and health care team to the procedures included in the study protocol (scheduled appointments, surveillance and transfusion strategies).
3. To determine the increase in hemoglobin levels and reticulocyte counts following a short-course of EPO plus supplemental Feraheme over a 1-4 week interval prior to the date of surgery vs. standard of care management in patients scheduled for CABG, valve, or CABG/valve surgery.
4. To assess differences in the proportion of patients receiving erythrocyte transfusions and number of blood products utilized (RBC, platelets and plasma) in the peri- and post-operative periods for those receiving a short-course of EPO plus supplemental Feraheme vs. standard of care management in patients scheduled for CABG, valve or CABG/valve surgery.
5. To determine the frequency and intensity of pre-defined clinical outcomes (mortality, major cardiac, renal, neurological events [associated with anemia] and infection) in the peri- and post-operative periods for those receiving a short-course of EPO plus Feraheme vs. standard of care management in patients scheduled for CABG, valve, or CABG/valve surgery.

Differences in hemoglobin levels and reticulocyte counts from baseline to the day of surgery and postop day (POD) 5, proportion of patients receiving transfusions and number of blood products utilized and the pre-defined clinical events will be assessed between the two groups. Each patient will be enrolled in the study up to 28 days before the day of surgery and for up to 30 days following the day of surgery. This pilot, feasibility study will enroll 50 subjects (25 per group). Both groups will have detailed clinical data and biological specimens collected.

Visits and Procedures:

* Screening: Patients undergoing cardiac surgery (CABG, valve, CABG/valve) with anemia will be identified in advance of their operations. Basic features of patient medical and surgical histories (i.e. age, gender, type of surgery) will be screened. If eligible for the study based on the inclusion/exclusion criteria, they will be consented into the study.
* Baseline Visit: Data on demographics, lab results, vital signs, medical history, current medications, height/weight will be reviewed and recorded. Randomization by computer will be done and the patient will receive the 1st dose of study drugs, as assigned, then monitored for any serious reactions (chest pain, dyspnea, seizures, severe headache, fever, nausea, vomiting, diarrhea, increase in BP). Control group patients with evidence of iron-deficiency by laboratory criteria will be advised to initiate supplementation with a non-prescription, over-the-counter oral iron preparation (ferrous sulfate 325 mg, three times a day is commonly used) to be taken until the planned surgical operation.
* Pre-op Visit: Patients will receive the 2nd dose of study drugs as assigned. Vital signs (heart rate, BP, oxygen saturation, temperature) will be recorded before and after drug administration, then monitored for any serious adverse events; SOC lab results; reticulocyte count, troponin, creatine kinase-myocardial band (CK-MB) samples will be collected.
* Day of Surgery: Patient vital signs (BP, electrocardiogram [EKG], etc) will be monitored as part of standard of care. Reticulocyte count, iron panel (includes transferrin, ferritin, total iron binding capacity, iron level) samples will be collected. SOC lab results, record of transfusions, estimated blood loss, adverse events will be monitored/recorded.
* POD 2: Troponin, CK-MB, Rotem (Rotational thromboelastometry) samples will be collected. Patients will receive study drug, as assigned, then monitored for serious events.
* POD 1-7: Vital signs (BP, EKG, etc) will be monitored; SOC lab results, record of transfusions, and adverse events will be monitored/recorded. Estimated blood loss will be recorded on POD 1 and 2 only.
* Other lab to be collected: POD 1 - reticulocyte count, iron panel, troponin, CK-MB; POD 2 - troponin, CK-MB, Rotem; POD 5 - reticulocyte count, iron panel, aspartate transaminase/alanine transaminase (AST/ALT); POD 7 - complete blood count (CBC), reticulocyte count, creatinine; POD 14 or discharge (whichever comes first) - CBC, creatinine.

Transfusion Strategy: Erythrocyte transfusion is permitted during cardiopulmonary bypass, during surgery and afterwards per protocol, when criteria is met. Red cell transfusions should be given one unit at a time with measurement of the pre- and post-transfusion hemoglobin levels along with physiologic parameters used to assess adequacy of organ perfusion. A consensus for transfusion thresholds was established among anesthesiologists, perfusionists and surgeons in our practice. The transfusion thresholds implemented in this protocol reflects our current "standard of care;" a threshold at which clinicians generally believe the benefits of erythrocyte transfusion outweigh the risks. Adherence to the transfusion strategy will be recorded by the research nurse and protocol deviations will be discussed with the attending physician of record and a member of the clinical research team. However, research staff will not order nor prohibit erythrocyte transfusions. This will be left to the discretion of the treating physician(s) if he/she deems it clinically necessary. Following randomization, patient's charts will be clearly labeled to indicate participation in the study protocol.

Surveillance Strategy: The decision to initiate and continue administering doses of EPO is based on evidence accrued from randomized controlled trials and clinical practice guidelines provided by multiple sub-specialty and international societies. Substantial heterogeneity exists in factors that could be included in a surveillance strategy to minimize the risk of a thrombotic event in this setting; with no one strategy proven to be superior. The surveillance strategy included in this protocol derives from, what we believe to be, the most current safety analyses of perioperative EPO use reflected in the literature. Implementing such surveillance methods are intended to minimize the possibly rare but potentially life-threatening adverse events. Risk factors considered in our surveillance strategy include: evidence of unstable angina or myocardial infarction, recent thrombotic event, hemoglobin levels associated with a higher risk of a myocardial event, excessive thrombocytosis or laboratory evidence of a hypercoagulable postoperative state. EPO dosing will be stratified based on patient risk (degree of perioperative anemia), type of procedure (CABG vs. valve) and laboratory data (hgb, Rotem). All doses will be given per surveillance guidelines.

Primary End Point: The primary objective is to assess the enrollment rate and adherence to the dosing protocol and surveillance strategies. We define successful adherence as adherence to dosing in more than 90% of patients for more than 90% of the doses deemed appropriate by the surveillance strategy. Secondary outcomes will include changes in hemoglobin levels and reticulocyte counts within the two groups from baseline to the day of surgery and POD 5, number of RBC units transfused, frequency of pre-specified clinical outcomes and incidence of adverse events in each of the study groups. Data from this pilot study will be used for the power analysis and design of the larger RCT.

Adverse events (AEs) are events that involve physiological, social, or psychological harm to subjects or risks of harm to additional subjects or others. AEs include expected and unexpected harmful effects, and unexpected risks of an interaction or an intervention. AEs may be caused by: the test article or test procedure, other aspects of the interaction or intervention, the subject's underlying condition, or the subject's concurrent standard treatment. AEs may be definitely related, probably related, possibly related, unlikely to be related, or definitely not related to the research. We will report all adverse events and other reportable incidences to the Institutional Review Board (IRB) per reporting guidelines. Any adverse event will be documented of that event including a description, subject number, date, outcome, and follow-up.

The primary safety endpoints of the study are the incidence of adverse events associated with the use of the study medications. These include: hypersensitivity (e.g. pruritis, rash, and urticaria), hypertension, hypotension, bleeding, nausea, vomiting, injection site pain, deep venous thrombosis or other thrombotic complications. Surveillance for these adverse events will be conducted by direct observation (during drug administration), daily bedside visits by the research nurse for the first 7 postoperative days, review of the patients medical record and listing any of these complications in the Society of Thoracic Surgery (STS) database. The definition of a stroke, myocardial infarction (MI), mesenteric artery occlusion or peripheral vascular event will be based on STS criteria. Any event resulting in death from time of initial drug administration to hospital discharge will be recorded.

The Principal Investigator, along with the Secondary Investigators, will be responsible for the monitoring, reviewing and analyses of study data. This will be done quarterly unless an issue requires immediate attention or if a recurrent pattern develops into a need for a more frequent review. An interim analysis will be done at 50% enrollment by the principal and secondary investigators.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 18 and 80 years old
* diagnosed with preoperative anemia, defined as hemoglobin <13.0 grams per deciliter (g/dL)
* scheduled for elective cardiac surgery (CABG, valve, or CABG/valve), including both first time and repeat procedures
* documented negative pregnancy test within 7 days prior to the procedure for females of child-bearing potential
* a written informed consent prior to any procedure, using a form that is approved by the UT Southwestern Institutional Review Board
* agreement to be compliant

Exclusion Criteria:

* uncontrolled hypertension (defined as systolic pressure greater than 180 millimeters of mercury (mmHg), diastolic pressure greater than 100mmHg, not adequately controlled by anti-hypertensive therapy at the time of procedure)
* current renal failure on dialysis or serum creatinine >3.0 milligrams per deciliter (mg/dL)
* unstable angina (defined by chest pain and EKG changes indicating ischemia at rest)
* thromboembolism within the past year
* current active primary or metastatic malignancy or history of myeloid malignancy
* seizures within the past year
* history of stroke within the last 6 months
* patients who have platelet count lower than 50,000 per cubic millimeter (mm3) or coagulation abnormality
* sepsis or bacteremia defined by positive blood culture
* patients who have known hypersensitivity to EPO or any of its components
* patients who have known hypersensitivity to Feraheme or any of its components
* patients who refuse blood transfusion, (i.e. Jehovah's Witnesses)
* pregnant or breast feeding
* patients who are unable to provide informed consent or who has inability to understand or corporate with study procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E. Greilich, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
All data and information collected during this study will be considered confidential and remains the sole property of UTSW Medical Center. Data may be shared with AMAG Pharmaceuticals, Inc., prior to any publications. All data used in the analysis and summary of this study will be anonymous, and without reference to specific subject names.

REFERENCES:
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EPO and Feraheme | Control
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPO and Feraheme | Control | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: # of Participants Who Adhered to the Study Protocol
Description: Successful adherence is defined as adhering to dosing in ≥90% of patients for ≥90% of the doses deemed appropriate by the surveillance strategy.
Time Frame: Preoperative 1st dose through Postoperative Day (POD) 2.
Measure: Count of Participants; unit: Participants
Arm/Group | EPO and Feraheme | Control
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

2. Secondary Outcome: Change From Baseline Hemoglobin Level Assessed at Different Time Points Within the 2 Arms.
Time Frame: Change from Baseline hemoglobin level to day of surgery (DOS), to POD 5.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dl)
Arm/Group | EPO and Feraheme | Control
Number analyzed (Participants) | 2 | 3
grams per deciliter (g/dl)
  Baseline hemoglobin level to DOS | 2.9 (1.1) | 3.33 (1.49)
  Baseline hemoglobin level to POD5 | 4.2 (0.2) | 2.2 (0.75)

3. Secondary Outcome: Change From Baseline Reticulocyte Count Assessed at Different Time Points Within the 2 Arms.
Time Frame: Change from Baseline reticulocyte count to DOS, to POD 5.
Population: Data were not collected for intervention group
Measure: Mean (Standard Deviation); unit: cells × 10^9/L
Arm/Group | EPO and Feraheme | Control
Number analyzed (Participants) | 0 | 3
cells × 10^9/L
  Baseline reticulocyte count to DOS |  | 0.43 (0.48)
  Baseline reticulocyte count to POD5 |  | 1.35 (0.95)

4. Secondary Outcome: Number of Blood Products Utilized Per Patient Receiving Erythrocyte Transfusions.
Description: Number of blood products utilized per patient receiving erythrocyte transfusions, including red blood cells, platelets and plasma.
Time Frame: Preoperative 1st dose through 30 days following surgery.
Measure: Mean (Standard Deviation); unit: blood product count
Arm/Group | EPO and Feraheme | Control
Number analyzed (Participants) | 2 | 3
blood product count | 2.5 (2.5) | 12.33 (2.36)

5. Secondary Outcome: Incidence of Pre-defined Clinical Events in Each of the Study Arms
Description: Incidence of mortality, major cardiac, renal, neurological events (associated with anemia) and infection. These events will include myocardial infarction, prolonged low-output state, encephalopathy, duration of mechanical ventilation, renal insufficiency,mortality and dialysis dependence at 30 days.
Time Frame: Preoperative 1st dose through 30 days following surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | EPO and Feraheme | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to discharge of the index surgery, including a 30 day follow-up. The average in-patient length of stay was 7.4 days in hospital.
Arm/Group | EPO and Feraheme | Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPO and Feraheme (N=2) | Control (N=3)
Cerebrovascular Accident (CVA) (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT02189889/Prot_SAP_000.pdf